CLINICAL TRIAL: NCT01957683
Title: A Multi-center Pilot Study Evaluating the Safety and Feasibility of the eCLIPs™ Family of Products for the Treatment of Unruptured Bifurcation Intracranial Aneurysms
Brief Title: Canadian eCLIPs™ Safety and Feasibility Study Protocol
Acronym: CESIS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: insufficient funds
Sponsor: Evasc Medical Systems Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS 13-003
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Intracranial Aneurysms
Keywords: intracranial aneurysm; bifurcation; wide-neck; saccular; endovascular treatment; coil embolization; stent; bare platinum
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Device: eCLIPs™ Family of Products

INTERVENTIONS:
Device: eCLIPs™ Family of Products — Safety and feasibility of the eCLIPs™ Family of Products for the treatment of unruptured bifurcation intracranial aneurysms
  Other Names: Bifurcation Remodeling Device; eCLIPs™ Microcatheter; eCLIPs™ Micro-Introducer; eCLIPs™ Detacher; eCLIPs™ Device; eCLIPs™ System; eCLIPs™ Products

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of the eCLIPs™ Family of Products for the treatment of unruptured intracranial bifurcation aneurysms in conjunction with embolization coils.

DETAILED DESCRIPTION:
With this other endoluminal stent/device implantation technique to treat intracranial aneurysms in conjunction with embolic coils, the neurovascular device is placed across the aneurysm neck, to act as a bridge to prevent coils from protruding into the parent artery. Stenting may allow to more safely achieve a higher packing density of coils. These effects may improve the rates of complete aneurysm occlusion and enhance the durability of the coiling treatment. The eCLIPs™ device manufactured by Evasc Medical Systems Corp. has a high density 'leaf' which is implanted across the bifurcation aneurysm neck and anchored in one of the branch arteries of the bifurcation and may provide improved bifurcation aneurysm treatment by allowing for a higher packing density of embolic coils implanted behind the eCLIPs™ device and the eCLIPs™ device in combination with embolic coils may reduce the recurrence/retreatment rate by increasing the rate of complete aneurysm occlusion.

ELIGIBILITY:
Inclusion

Only patients with the following characteristics are eligible for study entry:

1. Patient whose age is between 18 and 80 years old
2. Patient with an unruptured, saccular, intracranial aneurysm or recurrent aneurysm, which arises at a bifurcation and has a neck length of ≤ 6mm and aneurysm size of 5-35mm
3. Patient aneurysm arises at a bifurcation artery with at least one of the two branch artery vessels having a diameter between 2.0mm and 3.25mm
4. Patient understands the nature of the procedure and has the capacity to provide informed consent.
5. Patient is willing to have on-site 30- day, and 6-month, follow-up evaluations as per standard clinical practice.

Exclusion Criteria:

Patients with the following characteristics are not eligible for study entry:

1. Patient who presents with an intracranial mass or currently undergoing radiation therapy for carcinoma of the head or neck region.
2. Patient with an International Normalized Ratio (INR)≥ 1.5.
3. Patient with serum creatinine level ≥104 µmol/L at time of enrolment.
4. Patient with a platelet count ˂100x103 cells/mm3 or known platelet dysfunction at time of enrolment
5. Patient who has a known cardiac disorder, likely to be associated with cardioembolic symptoms such as AFIB (atrial fibrillation)
6. Patient with any condition which in the opinion of the treating physician would place the participant at a high risk of embolic stroke
7. Patient with known allergies to nickel-titanium metal
8. Patient with known allergies to aspirin, heparin, ticlopidine, or clopidogrel
9. Patient with a life threatening allergy to contrast (unless treatment for allergy is tolerated)
10. Patient with inappropriate anatomy as demonstrated by angiography due to severe intracranial vessel tortuosity or stenosis, or intracranial vasospasm not responsive to medical therapy.
11. Patient who is currently participating in another clinical research study.
12. Patient who has had a previous intracranial stenting procedure associated with the target aneurysm.
13. Patient who is unable to complete the required follow-up.
14. Patient who is pregnant or breastfeeding.
15. Patient who has participated in a drug study within the last 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
eCLIPs Bifurcation Remodelling System Technical Success | 24 hours
  The proportion of successful eCLIPs device implants at the target aneurysm.
No participant incurs a major stroke or death within 30 days or major territorial stroke or neurological death within 6 months. | 30 day-6 month
  A major stroke is defined as a new neurological event that persists for >24 hours and results in a 4 point increase in the NIHSS score compared to baseline or compared to any subsequent lower score.

OTHER OUTCOMES:
eCLIPs Microcatheter Technical Success | 24 hours
  The proportion of procedures where the eCLIPs Microcatheter is able to access the target vasculature and successfully deliver the eCLIPs device.
eCLIPs Micro-Introducer Technical Success | 24 hours
  The proportion of procedures where the eCLIPs Micro-Introducer successfully is used conjunction with the eCLIPs Microcatheter to assist in the delivery of the eCLIPs Microcatheter to the target aneurysm.
eCLIPs Detacher Technical Success | 24 hours
  The proportion of procedures where the eCLIPs Detacher is successfully used in conjunction with the eCLIPs Bifurcation Remodelling System to initiate detachment of the eCLIPs Device.
Measurement of aneurysm occlusion at 6 months | 6 months
  Successful aneurysm treatment with the eCLIPs™ device and embolic coils, as measured by aneurysm occlusion of ≥ 70% (Meyers grade of 2 or less) at 6 month follow up as measured by using standard medical practice radiographic imaging of either angiography, magnetic resonance angiography (MRA), or computed tomography angiography (CTA). The type of follow-up imaging is determined at the discretion of the treating physician.
Occurrence of unplanned aneurysm re-treatment within 6 months (endovascular or surgical repair). | 6 months
  As determined by the treating physician, where the patient has a ≤70% aneurysm occlusion corresponding to a Meyer's aneurysm occlusion grade of greater than 2 and the treating physician judges the need for the re-treatment.
Assessment of Device Migration at 6 months. | 6 months
  Radiographic images will be comparing post procedure device position to 6 months position to determine if migration has occurred. Imaging from each participant will be reviewed by an independent neuroradiologist who will be comparing baseline.
Assessment of artery stenosis at the device location at 6 months | 6 months
  Branch arteries will be measured at baseline and compared radiographically at 6 months post procedure per review by the Independent neuroradiologist.
Assessment of artery patency at the target aneurysm at 6 months | 6 months
  Patency will be assessed radiographically at 6 month follow up and assessed by an independent neuroradiologist.
Determination of percentage of screened patients who are eligible for the study | 24 hours
  The number of screened patients represents those patients reviewed by the investigator who have a known aneurysm and are considered for inclusion in the study. This represents the denominator of the proportion. The numerator will be the number of patients deemed eligible following the screening process.

CONTACTS AND LOCATIONS:
Overall Officials: Michael EB Kelly, PhD, MD, FRCSC, FACS, Principal Investigator — Royal University Hospital, Saskatoon, Saskatchewan
Locations (5):
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - Saint Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Hôpital de l'Enfant-Jésus, Québec